CLINICAL TRIAL: NCT07315737
Title: miRNAs Associated With Undescended and Retractile Testes
Brief Title: Could miRNAs be Used as Markers for Distinguishing Undescended Testicles From Retractile Testicles
Acronym: miRNA
Status: Completed | Type: Observational
Sponsor: Dr. Mevlüt Keleş (Other)
Responsible Party: Sponsor-Investigator, Dr. Mevlüt Keleş, Assistant professor, Ordu University
Organization: Ordu University (Other)
Other Study IDs: 2022/25; A-2109 (Other Grant/Funding Number: Ordu University Scientific Project Unit)
Record Dates: First submitted 2025-11-23; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: MIRAS; Testicular Abnominalies; Undescended Testes
Keywords: Cryptorchidism; Undescended testicle; Retractile testicle; miRNA; Infertility; Testicular cancer
MeSH Terms: conditions — Ataxia Neuropathy Spectrum; Cryptorchidism; Infertility; Testicular Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum samples collected for miRNA analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Undescended Testicle: Undescended testicle cases whose miRNA levels investigated
  Interventions: Diagnostic Test: miRNA
- Retractile testicle: Retractile testicle cases whose miRNA levels investigated
  Interventions: Diagnostic Test: miRNA
- Control: Healthy kids with testes in the scrotum whose miRNA levels investigated
  Interventions: Diagnostic Test: miRNA

INTERVENTIONS:
Diagnostic Test: miRNA — miR-34c , miR-210 , miR-449a levels investigated.

SUMMARY:
Background: Undescended testicles (UDTs) are common in male infants. Untreated UDT poses risks such as infertility (IF), testicular cancer (TC), and testicular torsion (TT). Retractile testicles (RTs) sporadically ascend from the scrotum. UDT requires early surgical correction, whereas RT requires only periodic follow-up. Differentiating these conditions is challenging, making clinical biomarkers potentially useful. The aim of our study was to examine the use of miRNAs, which are difficult to differentiate, as biomarkers in the differential diagnosis of UDT and RT.

Methods: This prospective study included 10 boys with UDT (operated), 9 with RT (followed), and 9 controls. Parent consent and serum samples were collected to evaluate miR-210, miR-34c, and miR-449a expression via real-time PCR. For group comparisons, one-way ANOVA was used for parametric data, and the Kruskal-Wallis test was used for nonparametric data, followed by the Dunn-Bonferroni correction for post hoc multiple comparisons. Spearman's rank correlation coefficient was used to analyse correlations. A p value < 0.05 was considered significant.

DETAILED DESCRIPTION:
1. Introduction Undescended testicles (UDTs) are the most common congenital male malformation, affecting 1.0-4.6% of term infants and up to 45% of preterm infants [1]. UDT can be congenital or acquired; spontaneous descent in congenital cases is rare after six months [2]. Untreated UDT beyond one year of age leads to interstitial fibrosis, degenerated spermatogenesis, and increased infertility risk [3-5]. Furthermore, untreated UDTs carry risks of testicular cancer (TC) and enhanced testicular torsion (TT). Early diagnosis and treatment are crucial to prevent these complications.

   Differentiating true underscended testicles (UDTs) from retractile testicles (RTs) is clinically challenging. True UDT involves a consistently empty scrotum, with testicles never descending. Conversely, RTs can spontaneously descend or be manually reduced, although they may reascend. Treatment for RT depends on the time spent outside the scrotum. Misdiagnosing UDT as RT risks delayed treatment and inevitable complications. Thus, reliable indicators for distinguishing UDTs and RT are crucial.

   MicroRNAs (miRNAs) are ~22-nucleotide noncoding RNAs that posttranscriptionally regulate gene expression [6]. MiRNAs are known to regulate spermatogenesis (SP), early embryonic development, sperm function, and fertilization in various species [7]. Given the expected SP disruption in true UDTs, the UDT-miRNA relationship has been explored. Studies have shown altered miRNA levels in UDT: miR-210 is upregulated [8], whereas miR-449a and miR-34c are downregulated [9-11]. Critically, data on miRNA changes in retractile testicle (RT) cases are currently lacking. Theoretically, the SP is not expected to be disrupted at RT. Thus, miRNA alterations, reflecting SP status, could differentiate RT from UDT, guiding surgical versus follow-up decisions. This study compared miRNA changes across UDT, RT, and normal control groups prospectively.
2. Materials and methods 2.1. Sample size This study is designed as a prospective controlled trial to compare miRNA changes across UDT, RT, and normal control groups. The sample size was determined via G*Power 3.1.9.6. A one-way ANOVA power analysis for miR-34c, which compared three groups, utilized an effect size (f=1.2955357) from a previous study [10]. To achieve 99% power and a 1% error rate, a total sample size of 24 was needed. To increase confidence, the study ultimately enrolled 30 patients, who were divided into three groups of 10.

2.2. Patient population Initially, 10 boys with undescended testicles (UDTs), 10 with retractile testicles (RTs), and 10 healthy volunteers (controls) from our urology clinic (dates between March 2022 and March 2023) were enrolled. However, one RT patient and one control patient were excluded because of parental refusal for blood sampling. Only palpable (unilateral or bilateral) UDT cases were included, excluding nonpalpable types. To ensure accurate RT diagnosis, initial physician examinations were performed in three positions (supine, semisupine, standing), followed by a 1-month parental examination (twice daily). Only RT patients whose testicles spent >50% of their time in the scrotum were included. The exclusion criteria also included prior inguinal/scrotal surgery, defective datasets, or unsuitable serum samples.

2.3. Collection of patient data and control samples Detailed patient histories, physical examinations, and routine biochemical tests were performed. UDT blood samples were collected presurgery to prevent misinterpretation. Blood from all the groups was collected in 5 mL biochemistry tubes and centrifuged at 3000 rpm for 10 minutes. The resulting particle-free serum was transferred to 1.5 mL tubes and stored at -80°C until analysis.

2.4. Validation of the expression levels of miR-210, miR-449a and miR-34c via real-time PCR Serum samples from the urology clinic were subjected to RNA isolation via the Quick-cfRNA™ Serum & Plasma Kit (Zymo Research). The extracted miRNA was reverse transcribed into cDNA via the miRNA All-In-One cDNA Synthesis Kit (ABMGood). cDNA quality and quantity were assessed spectrophotometrically with a BioSpec-nano instrument (Shimadzu) before real-time PCR. miRNA expression analysis was performed via a Rotor Gene Q (Qiagen) instrument. The levels of miR-210, miR-449a, and miR-34c were quantified with ready-to-use primers and BlasTaq™ 2X qPCR MasterMix (ABMGood).

2.5. Statistical analysis Data normality was assessed via the Shapiro-Wilk test, and variance equality was assessed via Levene's test. Descriptive statistics are presented as the means ± SDs for parametric data and medians (IQRs) and means (ranks) for nonparametric data. For group comparisons, one-way ANOVA was used for parametric data, and the Kruskal-Wallis test was used for nonparametric data, followed by the Dunn-Bonferroni correction for post hoc multiple comparisons. Spearman's rank correlation coefficient was used to analyse correlations. Statistical significance was set at p < 0.05.

miRNA expression was quantified via qRT-PCR via Ct (crossing point) values and normalized to RNU6B_13. Relative miRNA expression levels were compared among all groups via the 2-ΔCt method and calculated as 2Ct (target gene) - Ct (reference gene). All the statistical analyses were performed via IBM SPSS v28 (IBM Inc., Chicago, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* Palpable (unilateral or bilateral) undescended testis cases
* Retractile testis cases; physician examinations were performed in three positions (supine, semisupine, standing), followed by a 1-month parental examination (twice daily).
* Healty kids less than 18 years old with palpable two testes palpable in scrotum.

Exclusion Criteria:

* Prior inguinal/scrotal surgery
* Defective datasets
* Unsuitable serum samples

Ages: 3 Months to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — The study depends on undescended testicle which is a pathology related to male gender
Study Population: Control group: Healthy kids with both testes in scrotum. Undescended testis group: Kids with unilateral palpable undescended testis or bilateral palpable testes.
  Recractile testis group: Kids under monitorisation for unilateral retractile testis or bilateral retractile testes.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
miRNA levels | Within study enrollement
  2Ct (target gene) - Ct (reference gene)
miRNA changes | Rapid miRNA levels at study enrollement time.
  Differentiation of miRNA levels in three arms

CONTACTS AND LOCATIONS:
Overall Officials: Benli, Study Chair — Ordu University
Locations (1):
- Ordu University, Ordu, Altınordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pizzi G, Groppetti D, Brambilla E, Pecile A, Grieco V, Lecchi C. MicroRNA as epigenetic regulators of canine cryptorchidism. Res Vet Sci. 2023 Sep;162:104961. doi: 10.1016/j.rvsc.2023.104961. Epub 2023 Jul 20. PMID 37487386
- [Background] Kim EP, Shin JH, Kim WH, Kim GA. Integrated miRNA Changes in Canine Testis and Epididymis According to Age and Presence of Cryptorchidism. Animals (Basel). 2023 Apr 18;13(8):1390. doi: 10.3390/ani13081390. PMID 37106953
- [Background] Elias FM, Nishi MY, Sircili MHP, Bastista RL, Gomes NL, Ferrari MTM, Costa EMF, Denes FT, Mendonca BB, Domenice S. Elevated plasma miR-210 expression is associated with atypical genitalia in patients with 46,XY differences in sex development. Mol Genet Genomic Med. 2022 Dec;10(12):e2084. doi: 10.1002/mgg3.2084. Epub 2022 Nov 11. PMID 36369742
- [Background] Jia H, Ma T, Jia S, Ouyang Y. AKT3 and related molecules as potential biomarkers responsible for cryptorchidism and cryptorchidism-induced azoospermia. Transl Pediatr. 2021 Jul;10(7):1805-1817. doi: 10.21037/tp-21-31. PMID 34430428
- [Background] Yadav SK, Pandey A, Kumar L, Devi A, Kushwaha B, Vishvkarma R, Maikhuri JP, Rajender S, Gupta G. The thermo-sensitive gene expression signatures of spermatogenesis. Reprod Biol Endocrinol. 2018 Jun 2;16(1):56. doi: 10.1186/s12958-018-0372-8. PMID 29859541
- [Background] Procopio MS, de Avelar GF, Costa GMJ, Lacerda SMSN, Resende RR, de Franca LR. MicroRNAs in Sertoli cells: implications for spermatogenesis and fertility. Cell Tissue Res. 2017 Dec;370(3):335-346. doi: 10.1007/s00441-017-2667-z. Epub 2017 Aug 4. PMID 28779347
- [Background] Lian J, Zhang X, Tian H, Liang N, Wang Y, Liang C, Li X, Sun F. Altered microRNA expression in patients with non-obstructive azoospermia. Reprod Biol Endocrinol. 2009 Feb 11;7:13. doi: 10.1186/1477-7827-7-13. PMID 19210773
- [Background] Han H, Chen Q, Gao Y, Li J, Li W, Dang R, Lei C. Comparative Transcriptomics Analysis of Testicular miRNA from Cryptorchid and Normal Horses. Animals (Basel). 2020 Feb 21;10(2):338. doi: 10.3390/ani10020338. PMID 32098036
- [Background] Huang Z, Tang D, Gao J, Dou X, Cheng P, Peng D, Zhang Y, Mao J, Zhang L, Zhang X. miR-34c disrupts spermatogonial stem cell homeostasis in cryptorchid testes by targeting Nanos2. Reprod Biol Endocrinol. 2018 Oct 15;16(1):97. doi: 10.1186/s12958-018-0417-z. PMID 30322389
- [Background] Tang D, Huang Z, He X, Wu H, Peng D, Zhang L, Zhang X. Altered miRNA profile in testis of post-cryptorchidopexy patients with non-obstructive azoospermia. Reprod Biol Endocrinol. 2018 Aug 13;16(1):78. doi: 10.1186/s12958-018-0393-3. PMID 30103742
- [Background] Duan Z, Huang H, Sun F. The functional and predictive roles of miR-210 in cryptorchidism. Sci Rep. 2016 Aug 26;6:32265. doi: 10.1038/srep32265. PMID 27562222
- [Background] Lagos-Quintana M, Rauhut R, Meyer J, Borkhardt A, Tuschl T. New microRNAs from mouse and human. RNA. 2003 Feb;9(2):175-9. doi: 10.1261/rna.2146903. PMID 12554859
- [Background] Bartel DP. MicroRNAs: genomics, biogenesis, mechanism, and function. Cell. 2004 Jan 23;116(2):281-97. doi: 10.1016/s0092-8674(04)00045-5. PMID 14744438
- [Background] Park KH, Lee JH, Han JJ, Lee SD, Song SY. Histological evidences suggest recommending orchiopexy within the first year of life for children with unilateral inguinal cryptorchid testis. Int J Urol. 2007 Jul;14(7):616-21. doi: 10.1111/j.1442-2042.2007.01788.x. PMID 17645605
- [Background] Engeler DS, Hosli PO, John H, Bannwart F, Sulser T, Amin MB, Heitz PU, Hailemariam S. Early orchiopexy: prepubertal intratubular germ cell neoplasia and fertility outcome. Urology. 2000 Jul;56(1):144-8. doi: 10.1016/s0090-4295(00)00560-4. PMID 10869645
- [Background] Wenzler DL, Bloom DA, Park JM. What is the rate of spontaneous testicular descent in infants with cryptorchidism? J Urol. 2004 Feb;171(2 Pt 1):849-51. doi: 10.1097/01.ju.0000106100.21225.d7. PMID 14713841
- [Background] Radmayr C, Dogan HS, Hoebeke P, Kocvara R, Nijman R, Silay S, Stein R, Undre S, Tekgul S. Management of undescended testes: European Association of Urology/European Society for Paediatric Urology Guidelines. J Pediatr Urol. 2016 Dec;12(6):335-343. doi: 10.1016/j.jpurol.2016.07.014. Epub 2016 Sep 15. PMID 27687532
- [Background] Hadziselimovic F, Herzog B. The importance of both an early orchidopexy and germ cell maturation for fertility. Lancet. 2001 Oct 6;358(9288):1156-7. doi: 10.1016/S0140-6736(01)06274-2. PMID 11597673
- [Background] Moritoki Y, Hayashi Y, Mizuno K, Kamisawa H, Nishio H, Kurokawa S, Ugawa S, Kojima Y, Kohri K. Expression profiling of microRNA in cryptorchid testes: miR-135a contributes to the maintenance of spermatogonial stem cells by regulating FoxO1. J Urol. 2014 Apr;191(4):1174-80. doi: 10.1016/j.juro.2013.10.137. Epub 2013 Oct 31. PMID 24184258
- [Background] Jia H, Hao C. Exploring dysregulated miRNAs in cryptorchidism: a systematic review. J Int Med Res. 2021 Mar;49(3):300060521999950. doi: 10.1177/0300060521999950. PMID 33729892
- [Background] Lv W, Yu M, Su Y. miR-22-5p regulates the self-renewal of spermatogonial stem cells by targeting EZH2. Open Med (Wars). 2022 Mar 17;17(1):556-565. doi: 10.1515/med-2022-0429. eCollection 2022. PMID 35415251
- [Background] Garcia-Andrade F, Vigueras-Villasenor RM, Chavez-Saldana MD, Rojas-Castaneda JC, Bahena-Ocampo IU, Arechaga-Ocampo E, Diaz-Chavez J, Landero-Huerta DA. The Role of microRNAs in the Gonocyte Theory as Target of Malignancy: Looking for Potential Diagnostic Biomarkers. Int J Mol Sci. 2022 Sep 10;23(18):10526. doi: 10.3390/ijms231810526. PMID 36142439
- [Background] Dieckmann KP, Spiekermann M, Balks T, Ikogho R, Anheuser P, Wosniok W, Loening T, Bullerdiek J, Belge G. MicroRNA miR-371a-3p - A Novel Serum Biomarker of Testicular Germ Cell Tumors: Evidence for Specificity from Measurements in Testicular Vein Blood and in Neoplastic Hydrocele Fluid. Urol Int. 2016;97(1):76-83. doi: 10.1159/000444303. Epub 2016 Mar 19. PMID 26989896
- [Background] Condrat CE, Thompson DC, Barbu MG, Bugnar OL, Boboc A, Cretoiu D, Suciu N, Cretoiu SM, Voinea SC. miRNAs as Biomarkers in Disease: Latest Findings Regarding Their Role in Diagnosis and Prognosis. Cells. 2020 Jan 23;9(2):276. doi: 10.3390/cells9020276. PMID 31979244

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/37/NCT07315737/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/37/NCT07315737/ICF_001.pdf